CLINICAL TRIAL: NCT02081651
Title: Parmigiano-Reggiano Cheese as a Possible Strategy of Immunonutrition Able to Stimulate the Acquisition of Oral Tolerance in Childre With Cow's Milk Allergy
Brief Title: Parmigiano-Reggiano Cheese as a Possible Strategy to Acquire Oral Tolerance in Children With Cow's Milk Allergy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 272/13
Record Dates: First submitted 2014-02-27; First posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

ARMS (2):
- Parmigiano Reggiano cheese (Experimental): Children treated Parmigiano Reggiano cheese for 12 months
  Interventions: Dietary Supplement: Parmigiano Reggiano cheese
- Control subjects (No Intervention): Children with cow's milk allergy not assuming Parmigiano Reggiano cheese

INTERVENTIONS:
Dietary Supplement: Parmigiano Reggiano cheese
  Arms: Parmigiano Reggiano cheese

SUMMARY:
Cow's milk allergy is the most common food allergy in children. The scenery clinical and epidemiological of cow's milk allergy is significantly changed in the last decade. The severity of the clinical manifestations is still rising, and now cow's milk allergy has become the leading cause of hospitalization for food -induced anaphylaxis in our country. In addition, the overall prevalence of cow's milk allergy is increasing for a gradual reduction in the ability to acquire immunological tolerance to cow's milk protein in the first years of life. These mutations dictate the need to identify strategies to stimulate the acquisition of immunological tolerance in children affected by cow's milk allergy . The mechanisms of acquired immunological tolerance are not yet fully defined . The current view suggests the existence of a dynamic mechanism , consisting of various cellular compartments , which is set in a crucial environmental factors arising mainly from the diet and its effects on the intestinal microbiota. These acquisitions have contributed to the definition of a new concept in the field of human nutrition: immunonutrition. The immunonutrition is the ability, through the intake of specific nutrients on the immune system to interfere directly or indirectly through modulation of the composition and function of the intestinal microbiota. The proponent group has recently shown that it is possible to stimulate a more rapid acquisition of immunological tolerance in children affected by CMA through the administration of extensively hydrolysed casein containing the probiotic Lactobacillus rhamnosus GG (LGG) (Berni Canani et al. J Pediatr 2013) . Several lines of evidence suggest that this effect is induced by a combination of direct immunomodulatory action exerted by some small peptides derived from the beta - casein and the action of lactobacillus GG. It 's well known that the Lactobacillus GG is able to adjust the composition and functions of the microbiota in the child with CMA and directly adjust some immunological mechanisms involved in the pathogenesis of this condition. At the same time other groups have demonstrated the possibility that a high percentage of patients with IgE-mediated CMA is able to tolerate foods containing hydrolyzed cow's milk proteins with different processes. It has also been speculated that these strategies can facilitate the acquisition of immune tolerance in patients with cow's milk allergy. One of these foods is Parmigiano -Reggiano cheese, which is characterized by an ' extensive hydrolysis of the proteins in cow's milk , which degrade the caseins present and generate large amounts of peptides and free amino acids and by the presence of appreciable quantities of Lactobacillus GG in the samples to maturing higher . In a recent study it was shown that 58% of patients suffering from IgE-mediated CMA is able to tolerate a daily intake of normal amounts of this food , especially in the absence of a sensibilization to IgE specific to the beta lactoglobulin. These new findings allow us to hypothesize the use of Parmigiano REggiano cheese as a possible strategy immunonutrition can stimulate the acquisition of immune tolerance in patients with CMA .

ELIGIBILITY:
Inclusion Criteria:

-Children aged 3-10 years with cow's milk allergy

Exclusion Criteria:

* children aged less than 3 years or aged more than 10 years,
* concomitant chronic systemic diseases,
* active tubercolosis,
* autoimmune diseases,
* immunodeficiency,
* chronic inflammatory bowel disease,
* celiac disease,
* cystic fibrosis,
* metabolic diseases,
* malignancy,
* malformations of the gastrointestinal tract,
* suspected eosinophilic esophagitis or eosinophilic enterocolitis,
* suspected food-protien-induced enterocolitis syndrome,
* recent reaction to Parmigiano Reggiano cheese,
* pre/probiotic assumption

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who acquire immunological tolerance to cow's milk | After 12 months of intervention

SECONDARY OUTCOMES:
Rate of patients with positive skin prick test with Parmigiano Reggiano cheese | Enrollment and after 12 months of dietary treatment
Rate of patients able to tolerate the Parmigiano Reggiano cheese at enrollment | Enrollment
Differences in level of faecal butyrate after 12 months od treatment | After 12 months